CLINICAL TRIAL: NCT05158699
Title: The ESCRS EPICAT Study: Effectiveness of Periocular Drug Injection in CATaract Surgery
Brief Title: Effectiveness of Periocular Drug Injection in CATaract Surgery
Acronym: EPICAT
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Results of interim analysis: stop the trial due to one group being significantly different from the other three groups. Furthermore, shortage of study medication.
Sponsor: Luigi Rondas (Other)
Collaborators: European Society of Cataract and Refractive Surgeons (Other)
Responsible Party: Sponsor-Investigator, Luigi Rondas, Coordinating Investigator ESCRS EPICAT study, Academisch Ziekenhuis Maastricht
Organization: Academisch Ziekenhuis Maastricht (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NL72427.068.19; 2019-004890-21 (EudraCT Number)
Record Dates: First submitted 2021-11-21; First posted 2021-12-15 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-10

CONDITIONS: Macular Edema; Cystoid Macular Edema; Retinal Disease; Cataract; Lens Diseases; Eye Diseases
Keywords: Prevention
MeSH Terms: conditions — Macular Edema; Retinal Diseases; Cataract; Lens Diseases; Eye Diseases | interventions — bromfenac; Dexamethasone; Triamcinolone Acetonide; Triamcinolone

STUDY DESIGN:
Intervention Model Description: A block randomization procedure will be followed to acquire equal number of subjects in every treatment group. Patients are randomly allocated to 1 of 4 treatment groups in a 1:1:1:1 ratio. The various study centres will be taken into account during randomization.
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Masking will be achieved as much as possible. As there is an objective primary outcome, it will not be necessary to replace medicines by sham injections or placebo eye drops. Moreover, the ophthalmologist who performs the cataract surgery will not be blinded for treatment allocation of the subject. The study statistician, the data safety monitoring group, optometrists who perform the examinations (especially visual acuity) and observers who evaluate the examinations and OCTs will be masked when possible for treatment allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- topical bromfenac & dexamethasone (Active Comparator): bromfenac 0.09% eye drops twice daily starting two days before surgery and continuing 2 weeks postoperatively & dexamethasone 0.1% eye drops four times daily starting two days before surgery and continuing four times daily during the first postoperative week and one drop less per day every following week.
  Interventions: Drug: Bromfenac; Drug: Dexamethasone
- subconjunctival triamcinolone acetonide (Active Comparator): one subconjunctival injection of 10 mg triamcinolone acetonide during cataract surgery (TA, Triesence/Vistrec) in the inferotemporal quadrant, 6mm from the limbus.
  Interventions: Drug: Triamcinolone Acetonide
- intracameral ketorolac (Active Comparator): intracameral injection of ketorolac tromethamine solution during cataract surgery (Omidria). A 4ml vial of Omidria (ketorolac concentration 2.88mg/ml) is added to 500ml of the irrigation solution used during cataract surgery, resulting in a ketorolac concentration of 0.023mg/ml. At the end of the surgery, the anterior chamber will be filled with the ketorolac solution.
  Interventions: Drug: Ketorolac-Phenylephrine Ophthalmic 0.3%-1% Intraocular Solution
- subconjunctival triamcinolone acetonide & intracameral ketorolac (Active Comparator): one subconjunctival injection of 10 mg triamcinolone acetonide & intracameral injection of ketorolac tromethamine solution (Omidria; 0.023mg/mL) during cataract surgery.
  Interventions: Drug: Triamcinolone Acetonide; Drug: Ketorolac-Phenylephrine Ophthalmic 0.3%-1% Intraocular Solution

INTERVENTIONS:
Drug: Bromfenac — Bromfenac topical eye drops (Yellox)
  Other Names: Yellox; Product code: EU/1/11/692
  Arms: topical bromfenac & dexamethasone
Drug: Dexamethasone — Dexamethasone topical eye drops
  Other Names: Dexamethasone ophthalmic solution; Product code (NL): RVG 56003
  Arms: topical bromfenac & dexamethasone
Drug: Triamcinolone Acetonide — 0.25ml of 40mg/ml (10mg) triamcinolone acetonide (Triesence/Vistrec) will be injected subconjunctivally
  Other Names: Triesence or Vistrec; Product code (NL): RVG 106092
  Arms: subconjunctival triamcinolone acetonide; subconjunctival triamcinolone acetonide & intracameral ketorolac
Drug: Ketorolac-Phenylephrine Ophthalmic 0.3%-1% Intraocular Solution — Omidria is added to the irrigation fluid used during cataract surgery. At the end of surgery, the anterior chamber will be filled with the ketorolac solution.
  Other Names: Omidria
  Arms: intracameral ketorolac; subconjunctival triamcinolone acetonide & intracameral ketorolac

SUMMARY:
Cystoid macular edema (CME) is a major cause of suboptimal postoperative visual acuity after cataract surgery. Topical steroidal and nonsteroidal anti-inflammatory drugs (NSAIDs) are used to prevent CME. However, noncompliance with eye drops may compromise the effectiveness of treatment. Dropless periocular drug delivery during cataract surgery may improve the outcomes and cost-effectiveness of cataract surgery, and may alleviate the burden on homecare organizations.

DETAILED DESCRIPTION:
In a recent European multicentre study (PREvention of Macular EDema after cataract surgery; PREMED), it was demonstrated that the combination of topical corticosteroids and NSAIDs results in the lowest risk of developing CME after cataract surgery. However, noncompliance with eye drops may compromise the effectiveness of treatment. Noncompliance is often unintentional and related to forgetfulness or incorrect instillation, particularly in the elderly cataract surgery population.

The objective of this study is to evaluate the effectiveness of different treatments to prevent CME after cataract surgery, using either topical drugs (control group) or intra-/periocular injections (intervention groups).

The hypothesis of this study is that intra-/periocular anti-inflammatory drug delivery during cataract surgery is effective in preventing CME, with better health-related quality of life and improved cost-effectiveness compared to standard topical drug delivery.

The primary outcome measure is the change in central subfield mean macular thickness (CSMT) at 6 weeks postoperatively as compared to baseline. Secondary outcome measures are the incidence of CME; the incidence of clinically significant macular edema (CSME); mean corrected distance visual acuity (CDVA); para- and perifoveal thickness and total macular volume (TMV); intraocular pressure (IOP); anterior chamber inflammation; vision-related quality of life; and cost-effectiveness.

The design of this study is a European randomised controlled multicenter trial. The study population will consist of 808 patients aged 21 years or older who require cataract surgery in at least one eye. Patients with a foreseen increased risk of developing CME or ophthalmic disorders other than cataract will be excluded. Follow-up duration is 12 weeks. The study will be conducted over a period of 36 months.

ELIGIBILITY:
Inclusion Criteria:

* who are undergoing routine phacoemulsification (one eye per patient);
* who are 21 years or older;
* who should be able to communicate properly and understand instructions.
* willing and/or able to comply with the scheduled visits and other study procedures.

Exclusion Criteria:

* patients who already participated with their contralateral eye;
* combined surgery (e.g. combined phacoemulsification and trabeculectomy);
* patients with an increased risk of developing cystoid macular edema (CME) in the study eye (e.g. diabetes mellitus, previous retinal venous occlusion, or a history of uveitis, macular edema, epiretinal membrane, or previous retinal surgery);
* patients who developed CME after cataract surgery in the contralateral eye;
* patients with cystoid macular changes in the study eye at baseline;
* patients with an increased risk of developing perioperative complications (e.g. Fuchs' endothelial dystrophy);
* patients with permanent moderate visual impairment in the contralateral eye (decimal visual acuity less than 0.3);
* patients with a history of steroid induced IOP rise or glaucomatous visual field loss;
* patients using drugs that reduce or increase the risk of macular edema (e.g., periocular or intraocular corticosteroid, NSAID, or antivascular endothelial growth factor (VEGF) injection; topical corticosteroid or NSAID use; systemic corticosteroids (>= 20mg prednisolon), methotrexate, biologicals, or acetazolamide), or in the previous 4 months;
* patients with a contraindication for any of the investigated drugs;
* patients who are cardiovascular unstable;
* patients who have a history of hyperthyroidism.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 628 (Actual)
Dates: Start 2021-10-13 (Actual); Primary Completion 2024-08-13 (Actual); Study Completion 2024-08-13 (Actual)

PRIMARY OUTCOMES:
Change in central subfield mean macular thickness as a measurement of efficacy | Baseline, 6 weeks postoperatively
  The primary endpoint is the change in central subfield mean macular thickness in the 1 mm area (central subfield macular thickness, CSMT) as compared to baseline within the first 6 weeks postoperatively, measured using Optical Coherence Tomography (OCT)

SECONDARY OUTCOMES:
Change in central subfield mean macular thickness as a measurement of efficacy | Baseline, 12 weeks postoperatively
  Measured using OCT
No. of subjects developing clinically significant macular edema as a measurement of efficacy | Until 12 weeks postoperatively
  The occurrence of postoperative clinically significant macular edema (CSME) within 12 weeks postoperatively
Change in parafoveal retinal thickness in the central inner circle (1.0 - 3.0mm) as a measurement of efficacy | Baseline, 6 weeks and 12 weeks postoperatively
  Measured using OCT
Change in perifoveal retinal thickness in the central outer circle (3.0 - 6.0mm) as a measurement of efficacy | Baseline, 6 weeks and 12 weeks postoperatively
  Measured using OCT
Change in macular volume in the central 6.0mm area as a measurement of efficacy | Baseline, 6 weeks and 12 weeks postoperatively
  Measured using OCT
Change in corrected distance visual acuity (CDVA) as a measurement of efficacy | Baseline, 1 week, 6 weeks, and 12 weeks postoperatively
  CDVA measurements will be taken using Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity testing charts (logMAR)
Change in Intraocular pressure (IOP) as a measurement of safety | Baseline, 1 week, 6 weeks, and 12 weeks postoperatively
  IOP (in mmHg) will be measured by Goldmann applanation tonometry (preferred), Non-Contact Tonometry, or iCare tonometry
Anterior chamber inflammation as a measurement of safety | Baseline, 1 week , 6 weeks, and 12 weeks postoperatively
  Grading will be performed using the classification of the "Standardization of Uveitis Nomenclature" (SUN) working group using a 2mm long and 1mm wide slit beam:
  1. grading aqueous cells between grade 0 [<1cell, best outcome] up to grade +4 [>50 cells, worse outcome]
  2. grading aqueous flare between grade 0 [none detectable] up to +4 [intense aqeous flare or fibrinous exudate] Higher grade scores mean a worse outcome.
No. of subjects with Adverse Events as a measurement of safety and tolerability | Until 12 weeks postoperatively
  An adverse event (AE) is defined as any undesirable experience occurring to a subject during the study, whether or not considered related to the investigational product. All adverse events reported spontaneously by the subject or observed by the principal investigator or his staff will be recorded.
  Most frequently reported adverse events which might occur while using the study medication: abnormal sensation in the eye, pain or irritation, redness or headache while using eye drops; increased IOP and masking of infections while using corticosteroids; abnormal sensation in the eye, pain or irritation, conjunctival hyperaemia, inflammation and corneal edema after intracameral injection with phenylephrine/ketorolac.
Patient reported outcome measures (PROMs): NEI VFQ-25 | Baseline and 12 weeks postoperatively
  Patient satisfaction and vision-specific quality of life as measured by National Eye Institute Visual Function Questionnaire (NEI VFQ-25). From 25 questions, the original numeric values given (1-10) are converted to a 0 to 100 scale, so that the scores are set between 0 points (worst outcome) and 100 points (best outcome).
Patient reported outcome measures (PROMs): Catquest-9SF | Baseline and 12 weeks postoperatively
  Patient satisfaction and vision-specific quality of life as measured by the Catquest-9SF questionnaire. The possible range in Catquest scores are -3.94 (no difficulties) to +3.52 (great difficulties).
Patient reported outcome measures (PROMs): HUI3 | Baseline and 12 weeks postoperatively
  Health-related quality of life as measured by HUI3 (Health Utility Index Mark 3) questionnaire. The HUI3 questionnaire consists of 8 attributes, including vision, hearing, speech, ambulation, dexterity, emotion, cognition, and pain. For each attribute, the HUI3 questionnaire provides utility (preference) scores on a generic scale where dead = 0.00 and perfect health = 1.00.
Patient reported outcome measures (PROMs): EQ-5D-5L | Baseline and 12 weeks postoperatively
  Health-related quality of life as measured by the 5-level EQ-5D version (EQ-5D-5L) questionnaire. The EQ-5D-5L consists of the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS).
  1. The EQ-5D descriptive system results in a number between 1 (best) and 5 (worse) that expresses the level selected for that dimension.
  2. The EQ VAS indicates the general health status with 0 indicating the worst and 100 indicating the best health status.
Quality Adjusted Life Years (QALYs) | Baseline until 12 weeks postoperatively
  Calculated based on generic health-related quality of life, using the EQ-5D-5L and HUI-3 questionnaires
Costs per patient | Baseline until 12 weeks postoperatively
  Cost per patient, including valuation of resource use by using the Dutch guidelines for cost-analyses or cost prices provided by the medical center.
Incremental cost-effectiveness ratios (ICERs): QALY | Baseline until 12 weeks postoperatively
  Evaluation of cost-effectiveness by using calculated costs per quality-adjusted life years (QALYs)
Incremental cost-effectiveness ratios (ICERs): NEI VFQ-25 | Baseline until 12 weeks postoperatively
  Calculated costs per clinically improved patient on the NEI VFQ-25 questionnaire
Incremental cost-effectiveness ratios (ICERs): Catquest | Baseline until 12 weeks postoperatively
  Calculated costs per clinically improved patient on the Catquest questionnaire
Incremental cost-effectiveness ratios (ICERs): Visual acuity | Baseline until 12 weeks postoperatively
  Calculated costs per patient with clinical improvement in (un)corrected distance visual acuity
Budget impact | Baseline until 12 weeks postoperatively
  Reported as a difference in costs. Different scenario's will be compared to investigate the impact of various levels of implementation (e.g. 25%, 50%, 75% of eligible patients).

CONTACTS AND LOCATIONS:
Overall Officials: Nienke Visser, Dr., Principal Investigator — Universiteitskliniek voor Oogheelkunde Maastricht UMC+
Locations (10):
- Austria (2):
  - Hospital of the Brothers of Saint John of God, Vienna
  - Vienna Institute for Research in Ocular Surgery, Hanusch Krankenhaus, Vienna
- Goethe University, Frankfurt am Main, Germany
- Netherlands (6):
  - Amphia, Breda
  - Deventer Ziekenhuis, Deventer
  - Zuyderland Medisch Centrum, Heerlen
  - University Eye Clinic Maastricht UMC+, Maastricht
  - Canisius Wilhelmina Ziekenhuis Nijmegen, Nijmegen
  - Elisabeth-Twee Steden Ziekenhuis, locatie Elisabeth, Tilburg
- University Hospital Coimbra, Coimbra, Portugal

IPD SHARING:
Plan to Share IPD: No